CLINICAL TRIAL: NCT05630586
Title: The Safety and Efficacy of Acute Subcutaneous Administration of Semaglutide in Non-diabetic Patients With Acute Ischemic Stroke: A Multicentre, Phase 2, Prospective, Randomized, Open-label, Blinded Endpoint Trial
Brief Title: Acute Subcutaneous SemaglutidE in Acute Ischemic sTroke
Acronym: ASSET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); Glostrup University Hospital, Copenhagen (Other); Odense University Hospital (Other); Herning Hospital (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASSET; EUCT number: 2022-501072-25-02 (Other: European Medicines Agency (EMA))
Record Dates: First submitted 2022-11-01; First posted 2022-11-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — semaglutide; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide 0.5 mg (Active Comparator): Inj. Semaglutide 0.5 mg s.c., 0.5 mg per week for 4 weeks
  + standard care
  Interventions: Drug: Semaglutide; Other: Standard care
- Control (Other): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Semaglutide — Subcutaneous Semaglutide, 0.5 mg weekly for 4 weeks. First dose given at inclusion.
  Other Names: Ozempic
  Arms: Semaglutide 0.5 mg
Other: Standard care — Treatment according to Danish national clinical guidelines on stroke treatment, including reperfusion therapy if eligible.

SUMMARY:
Can Semaglutide help reduce the damage caused by a stroke? ASSET trial is a national, multicenter, clinical trial, investigating the safety and efficacy of Semaglutide in non-diabetic patients with acute ischemic stroke.

Stroke is a worldwide leading cause of long-term disability and death. In the most common type of stroke (ischemic stroke), a blood clot obstructs an artery in the brain, and thereby prevents oxygenated blood from reaching an area of the brain. Brain cells are particularly vulnerable to the lack of oxygen. In the areas most severely affected by a stroke, brain cells die after 5 minutes. As more time pass, the affected area expands, and more brain cells perish. Today, efficient treatments aiming at reestablishing the flow of blood by either breaking down the blood clot (thrombolysis) or removing the clot (thrombektomi) are used. However, a significant amount of patients undergoing succesful treamtent, still suffer permanent disability following an ischemic stroke.

Semaglutide mimics a naturally occurring hormone (glucagon-like peptide-1) and is currently used to treat diabetes and obesity. However, semaglutide has also been shown to possess neuroprotective abilities in recent animal studies, where it reduced the damage caused by ischemic stroke in rats. This study sets out to investigate if it's possible to utilize Semaglutide, to increase the resilience of brain cells in patients with an acute ischemic stroke, with the aim of bettering their outcome.

The participants consist of non-diabetic patients with acute ischemic stroke, who will be randomized to:

* Treatment with subcutaneous Semaglutide, or
* No additional treatment (control group)

Both groups will be treated according to the standard national guidelies for acute ischemic stroke.

The two groups will then be compared to see, if patients in the group treated with Semaglutide are less impacted by their stroke.

DETAILED DESCRIPTION:
For detailed project description, please refer to the full trial information at the Clinical Trials Information System (see 'More information' below for link).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients (≥ 18 years) at the time of signed informed consent/proxy consent
* Acute ischemic stroke with disabling neurological deficits (defined as an impairment of one or more of the following: language, motor function, cognition, gaze, vision, neglect, or ataxia)
* Onset/last seen well to randomization < 4.5 hours
* None to moderate disability in daily living before symptom onset (pre-stroke modified Rankin Scale 0-3)

Exclusion Criteria:

* Diabetes (known) or plasma/point of care test-glucose >11.1 mmol/L at admission
* BMI< 22
* History of pancreatitis, medullary thyroid carcinoma
* Predisposition or known Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* Short remaining life expectancy (< 12months) and/or severe neurodegenerative disease
* Pregnancy or planned pregnancy within 12 months or breastfeeding
* Renal impairment measured as estimated glomerular filtration rate (eGFR) value of <30 mL/min/1.73 m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Modified Ranking Scale | 90 (+/- 14) days
  A shift towards better functional outcomes in the distribution of the modified Ranking Scale (mRS)

SECONDARY OUTCOMES:
Serious Adverse Events and/or Serious Unexpected Serious Adverse Events | 90 days
  Proportion of patients with Serious Adverse Events (SAE) and/or Serious Unexpected Serious Adverse Events (SUSAR) within 90 days of randomization
90-day mortality | 90 days
One-year mortality | 1 year
Predefined SAEs | 1 year
  Frequency of predefined serious adverse events
Excellent functional outcome at 90 days | 90 (+/- 14) days
  mRS score of 0-1
MACCE and recurrent ischemic events, 90 days | 90 days
  Major Adverse Cardiac and Cerebral Events (MACCE) and recurrent ischemic events based on registry data at 3 months in AIS patients
MACCE and recurrent ischemic events, 12 months | 12 months
  Major Adverse Cardiac and Cerebral Events (MACCE) and recurrent ischemic events based on registry data at 12 months in AIS patients
Stroke recurrence at 12 months in patients with a stroke due to small vessel disease | 12 months
Early neurological improvement | 24 (+/- 8) hours
  NIHSS_24hour - NIHSS_baseline (NIHSS National Institutes of Health Stroke Scale)
Change in body weight (kg) | 90 (+/- 14) days
  90 days - baseline
Change in fasting plasma glucose | 90 (+/- 14) days
  90 days - baseline
Change in body mass index (BMI) | 90 (+/- 14) days
  90 days - baseline
Change in waist circumference | 90 (+/- 14) days
  90 days - baseline
Difference in HbA1c | 90 (+/- 14) days
  90 days - baseline
Diabetes diagnosis and/or antidiabetic medication | 12 months
  Diagnosed with and/or started antidiabetic medication within 1 year of enrollment
Blood pressure, 90 days | 90 (+/- 14) days
  Systolic and diastolic blood pressure (90 days BP - discharge BP)

OTHER OUTCOMES:
Patient reported outcome: Quality of Life (QoL) | 90 (+/- 14) days
  European Quality of Life - 5 Dimension (EQ5D), 90 days - baseline
Patient reported outcome: Major Depression Inventory (MDI) | 90 (+/- 14) days
  Change in MDI (90 days - baseline)
Patient reported outcome: SSQOL-DK | 90 (+/- 14) days
  Difference in Stroke Specific Quality of Life Scale (SSQOL-DK, 90 days)
Patient reported outcome: Activities of daily living | 90 (+/- 14) days
  Difference in activities of daily living - Multi Data Set -Home Care (MDS-HC,90 days)
Sub-study: 24-hour infarct growth | 24 (+/-8) hours
  Infarct growth on diffusion-weigthed magnetic resonance imaging (DWI-MRI). Aarhus University Hospital (AUH) only
Sub-study: Acute and long-term platelet inhibition in Semaglutide treated patients | 90 (+/- 14) days
  AUH only
Sub-study: The effect of semaglutide in non-diabetic stroke patients on insulin, c-peptide, glucagon and 3-hydroxybuturate levels | 90 (+/- 14) days
  AUH only
Sub-study: The effect of semaglutide in non-diabetic stroke patients on leptin, ghrelin, cholecystokinin (CCK) and gastric inhibitory polypeptide (GIP) | 90 (+/- 14) days
  AUH only

CONTACTS AND LOCATIONS:
Overall Officials: Claus Z Simonsen, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Trial informaion on CTIS (Clinical Trials Information System), European Medicinal Agency — https://euclinicaltrials.eu/view-clinical-trial?p_p_id=emactview_WAR_emactpublicportlet&p_p_lifecycle=0&p_p_state=normal&p_p_mode=view&p_p_col_id=column-1&p_p_col_count=1&_emactview_WAR_emactpublicportlet_number=2022-501072-25-02&_emactview_WAR_emactpublicportlet__facesViewIdRender=%2FWEB-INF%2Fviews%2Fview%2Ftabs%2Fsummary.xhtml